CLINICAL TRIAL: NCT05532371
Title: Is Aerobic and Dual-task Training Combination the Most Effective Exercise Combination to Improve the Cognitive Status and Physical Function in Older Adults With Mild Cognitive Decline
Brief Title: The Effect of Exercise on Cognitive Status in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ismail Uysal, İsmail Uysal, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gazi University
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Older People

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise training combined with lower limb strengthening group (AG) (Experimental): Aerobic exercise training combined with lower limb strengthening.
  Interventions: Other: Aerobic exercise training combined with lower limb strengthening
- Dual-task training combined with lower limb strengthening group (DG) (Experimental): Dual-task training combined with lower limb strengthening.
  Interventions: Other: Dual-task training combined with lower limb strengthening group (DG)
- Aerobic exercise training combined with dual-task training and lower limb strengthening group (ADG) (Experimental): Aerobic exercise training combined with dual-task training and lower limb strengthening.
  Interventions: Other: Aerobic exercise training combined with dual-task training and lower limb strengthening
- Only lower limb strengthening group (CG) (Active Comparator): Only lower limb strengthening.
  Interventions: Other: Only lower limb strengthening group (CG)

INTERVENTIONS:
Other: Aerobic exercise training combined with lower limb strengthening — The participants performed aerobic exercise training and lower limb strengthening during this intervention.
  Arms: Aerobic exercise training combined with lower limb strengthening group (AG)
Other: Dual-task training combined with lower limb strengthening group (DG) — The participants performed dual-task training combined with lower limb strengthening during this intervention.
  Arms: Dual-task training combined with lower limb strengthening group (DG)
Other: Aerobic exercise training combined with dual-task training and lower limb strengthening — The participants performed aerobic exercise training combined with dual-task training and lower limb strengthening during this intervention.
  Arms: Aerobic exercise training combined with dual-task training and lower limb strengthening group (ADG)
Other: Only lower limb strengthening group (CG) — The participants performed only lower limb strengthening group during this intervention.
  Arms: Only lower limb strengthening group (CG)

SUMMARY:
The purpose of the study is to demonstrate the effectiveness of the different combinations of exercises on the cognitive status of older adults with cognitive decline.

DETAILED DESCRIPTION:
This study is planned to examine the effects of combined exercise on cognitive status, lower extremity muscle strength, mobility, physical performance, mood and quality of life in older adults with Mild Cognitive Impairment. Aerobic exercise training and lower limb (extremity) strengthening exercises were applied to the first group, dual-task training and lower limb strengthening exercises were applied to the second group, and aerobic exercise training, dual-task training and lower limb strengthening exercises were applied to the third group.

ELIGIBILITY:
Inclusion Criteria:

* Not had a fall in the last six months.
* Older adults with an mini mental state examination score between18-23.
* Age ≥ 65years.

Exclusion Criteria:

* having central nervous system pathology that will affect balance
* diagnosed with vestibular pathology,
* having deformities in the waist, hip, and knee joints,
* having lower extremity amputation,
* with lower extremity operation history,
* malignancy affecting the lower extremity,
* having moderate and severe congenital heart disease, coronary heart disease and cerebrovascular disease,
* participants who cannot cooperate,
* participants who use an assistive walking device,
* participants having vision problems.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 12 weeks
  Cognitive status examination is applied with a simple test called "Mini-Mental State Examination".
Commander Power Track 2 Manual Tester | 12 weeks
  Muscle strength strength is carried out with "Commander Power Track 2 Manual Tester".
Timed Up and Go Test | 12 weeks
  Functional mobility is evaluated by Timed Up and Go Test.
Single Leg Stance Test | 12 weeks
  Static balance is evaluated by Single Leg Stance Test
Activities-specific Balance Confidence Scale | 12 weeks
  Balance Confidence is evaluated by Activities-specific Balance Confidence Scale.
Six-Minute Walk Test | 12 weeks
  Exercise capacity is evaluated by Six-Minute Walk Test.
Short Physical Performance Battery | 12 weeks
  Physical performance is evaluated by Short Physical Performance Battery.
Hamilton Depression Rating Scale | 12 weeks
  Emotional status is evaluated by Hamilton Depression Rating Scale
World Health Organization Quality of Life-Old module | 12 weeks
  Quality of life is evaluated by World Health Organization Quality of Life-Old module

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Uysal, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No